CLINICAL TRIAL: NCT02663570
Title: Effects of 6 Months of Melatonin Treatment on Clinical, Endocrine ed Metabolic Features in Women Affected by PCOS
Brief Title: Effects of Melatonin in PCOS Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Rosanna Apa, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Melatonina15
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Melatonin

ARMS (1):
- open (Experimental): therapy with melatonin 2 mg daily for six months
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin

SUMMARY:
The aim of our study is to investigate the effects of a treatment with melatonin on clinical, endocrine and metabolic features in women affected by PCOS. The study group included 40 patients treatend with 2 mg of melatonin daily for six months. Menstrual pattern, anthropometric parameters, hirsutism score, ultrasound ovarian volume and antral follicular count, an oral glucose tollerance test and hormonal assays are evaluated before and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS in accordance with Rotterdam criteria

Exclusion Criteria:

* pregnancy
* past history of cardiovascular diseases
* diabetes mellitus (or impaired glucose tolerance as determined by a standard 75 gr oral glucose tolerance test)
* hypertension
* significant liver or renal impairment
* other hormonal dysfunction (hypothalamic, pituitary, thiroidal or adrenal)
* neoplasms

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of cycles in six months of therapy | 6 months

SECONDARY OUTCOMES:
hirsutism score | 6 months
  Ferriman Gallwey score
testosterone levels | 6 months
insulin levels | 6 months
total cholesterol | 6 months
HDL cholesterol | 6 months
LDL cholesterol | 6 months
tryglycerides | 6 months
androstenedione levels | 6 months
free androgen index | 6 months
AMH levels | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic university of Sacred Heart, Rome, Rome, Italy